CLINICAL TRIAL: NCT00964288
Title: A Double Blind, Double Dummy, Placebo Controlled Cross Over Study With a Positive Control to Investigate the Effect of a GSK Drug on Electrical Hyperalgesia and Threshold Tracking in Healthy Subjects
Brief Title: Effect of GSK1014802 on Electrical Hyperalgesia and Threshold Tracking in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: During treatment session 3, a subject had a pattern of AEs of severe intensity, suggestive of brainstem toxicity/encephalopathy during lidocaine/saline infusion
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111676; NP111676
Record Dates: First submitted 2009-07-23; First posted 2009-08-24 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Pain, Neuropathic; Neuropathic Pain
Keywords: electrical hyperalgesia; threshold tracking; pain
MeSH Terms: conditions — Neuralgia; Pain | interventions — vixotrigine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Period 1 (Other)
  Interventions: Drug: GSK1014802 low dose; Drug: Lidocaine; Drug: GSK1014802 high dose; Drug: Placebo
- Period 2 (Other)
  Interventions: Drug: GSK1014802 low dose; Drug: Lidocaine; Drug: GSK1014802 high dose; Drug: Placebo
- Period 3 (Other)
  Interventions: Drug: GSK1014802 low dose; Drug: Lidocaine; Drug: GSK1014802 high dose; Drug: Placebo
- Period 4 (Other)
  Interventions: Drug: GSK1014802 low dose; Drug: Lidocaine; Drug: GSK1014802 high dose; Drug: Placebo

INTERVENTIONS:
Drug: GSK1014802 low dose — oral tablet
  Other Names: BIIB074 and CNV1014802
Drug: Lidocaine — positive control
Drug: GSK1014802 high dose — oral tablet
  Other Names: BIIB074 and CNV1014802
Drug: Placebo — To match GSK drug and positive control

SUMMARY:
This study is being conducted to assess the effects of GSK1014802 and a positive control, lidocaine, on tests of peripheral nerve excitability. This will be a double blind, placebo controlled, 4-period cross over study. Approximately 20 subjects will be randomised to one of two doses of a GSK1014802, lidocaine and placebo with at least 2 weeks between sessions. A follow-up will occur 7-15 days after the last dose.

During treatment session 3 on the 6th October 2009, one subject had a pattern of AEs of severe intensity, suggestive of brain stem toxicity / encephalopathy during the lidocaine/saline infusion period. Although recognised in the literature when lidocaine was used in patients for treatment of pain, these AEs were unusual in studies in healthy subjects. The study was suspended to allow re-evaluation of the risk:benefit balance of lidocaine/saline infusion in healthy subjects in this study. It was decided that continuation of the use of lidocaine (positive control) would risk the safety of subjects. Continuation without the positive control was not possible as it would compromise the scientific integrity of the design.

DETAILED DESCRIPTION:
This study, previously posted by GlaxoSmithKline (GSK), was transitioned to Convergence Pharmaceuticals, Ltd., which spun off from GSK. Convergence Pharmaceuticals, Ltd., has now been acquired by Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 55 years of age inclusive.
* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN
* Healthy as determined by a responsible and experienced physician.
* Male subjects must agree to use one of the contraception methods requested.
* Body weight greater than or equal to 50 kg, BMI ≤29.9kg/m2
* Capable of giving written informed consent.
* QTcB or QTcF < 450 msec.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Heart block, bundle branch block, hemi-block, evidence of accessory cardiac conduction pathways, long pauses >2 s or other cardiac conduction abnormalities or cardiac arrhythmias on 12-lead ECG or 24 h Holter at screening.
* History of regular excessive alcohol consumption within 6 months of the study.
* The subject has participated in a clinical trial and has received an investigational product within 90 days o fthe strat of this study.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Subjects with a history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Average daily caffeine intake equivalent to > 4 cups of coffee or > 6 cups of tea.
* Current or past history of symptomatic orthostatic hypotension or history of vasovagal episode(s).
* Subjects with systolic blood pressure persistently above 140 mmHg and/or diastolic blood pressure persistently above 90 mmHg.
* History of known or suspected seizures, including infantile febrile, unexplained significant and recent loss of consciousness or history of significant head trauma with loss of consciousness or a family history (first degree relative) of epilepsy or seizures (fits).
* The subject has a history of chronic pain before screening.
* The subject has used any topical steroid in the previous 30 days if, in the opinion of the investigator this is likely to interfere with study assessments.
* The subject has used any topical capsaicin preparations on the forearms in the previous 30 days.
* The subject suffers from eczema, psoriasis or any other acute or chronic dermatological problem if, in the opinion of the investigator this is likely to interfere with study assessments
* The subject suffers from tinnitus, or has done in the past 3 months.
* Suffers from skin infection or inflammation of the forearm, or has other arm skin irregularities that may in the opinion of the investigator interfere with study assessments.
* Needle phobic.
* The subject does not produce an area of allodynia or hyperalgesia to the electrical hyperalgesia model during the screening session.
* The subject is unable to tolerate the electrical hyperalgesia model or threshold tracking, including anxiety or atypical response to the stimulation.
* Any history of suicidal behaviour or any suicidal ideation of type 4 or 5 on the C-SSRS in the last month.
* Poor veins that would be estimated not to be suitable by a physician for repeated cannulation in both arms.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-11-30 (Actual)

PRIMARY OUTCOMES:
To determine the effect of single oral doses of GSK1014802 on area of flare evoked by cutaneous electrical stimulation. | 16 weeks

SECONDARY OUTCOMES:
To determine the effect of single oral doses of GSK1014802 and a single i.v. infusion of lidocaine on tests of nerve excitability | 16 weeks
To further investigate the safety and tolerability of single oral doses of GSK1014802 | 16 weeks
To assess relationships between GSK1014802 pharmacokinetics and pharmacodynamic endpoints. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Medical Director, Study Director — Biogen